CLINICAL TRIAL: NCT05750043
Title: Effect of Onchocerciasis Elimination Measures on the Incidence of Epilepsy in Maridi, South Sudan, a Three-year Prospective Study
Brief Title: Effect of Onchocerciasis Elimination Measures on the Incidence of Epilepsy in Maridi, South Sudan
Acronym: OAEMaridi
Status: Completed | Type: Observational
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Amref Health Africa (Other)
Responsible Party: Principal Investigator, Robert Colebunders, Professor, Universiteit Antwerpen
Other Study IDs: Project Code AID 011898
Record Dates: First submitted 2023-02-19; First posted 2023-03-01 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Onchocerciasis; Epilepsy
MeSH Terms: conditions — Onchocerciasis; Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Population of selected villages in Maridi county: A total of 2,511 households containing 17,652 individuals were visited in 2018, and 2,254 households containing 14,402 individuals in 2022.
  Interventions: Drug: bi-annual CDTI

INTERVENTIONS:
Drug: bi-annual CDTI — bi-annual community directed treatment with ivermectin (CDTI) and community-based "slash and clear" vector control intervention
  Other Names: "slash and clear" vector control intervention

SUMMARY:
For the first time using a prospective design, a study confirms the results of previous retrospective studies, which found that strengthening onchocerciasis elimination efforts decreases the incidence of epilepsy, including nodding syndrome. Therefore, this study confirms the solid epidemiological link between onchocerciasis and epilepsy.

This study also shows that a community-based "Slash and Clear" vector control method can effectively decrease blackfly biting rates and potentially decrease onchocerciasis transmission.

Moreover, this study shows that epilepsy is a major cause of death in onchocerciasis endemic areas with high ongoing transmission.

DETAILED DESCRIPTION:
Background High onchocerciasis transmission predisposes communities in endemic areas to a high epilepsy burden. The 4·4% (95%CI:4·1-4·7%) epilepsy prevalence documented in 2018 in Maridi, South Sudan, motivated the strengthening of onchocerciasis elimination measures. We evaluated the effect of these interventions on the incidence of epilepsy, including nodding syndrome (NS).

Methods Annual community-directed treatment with ivermectin (CDTi) was implemented in 2019, temporarily interrupted in 2020 and reimplemented biannually in 2021. Additionally, a community-based "Slash and Clear" vector control method was initiated in 2019 at the Maridi dam. A two-stage house-to-house survey was conducted before (2018) and after (2022) implementing the interventions, consisting of initial screening by community workers to detect suspected cases of epilepsy, followed by confirmation of the diagnosis by a trained clinician.

Finding Overall, 17,652 and 14,402 individuals participated in the pre- and post-intervention surveys, respectively. The epilepsy incidence decreased from 313·0 (95% confidence intervals (CI):273·7-357·7) to 34·7 (95%CI:17·6-66·1) per 100,000 person-years. Similarly, the incidence of NS decreased from 120·4 (95%CI:96·7-149·6) to 10·4 (95%CI:2·7-33·2) per 100,000 person-years. Despite biannual CDTi, only 56·6% of the population took ivermectin in 2021. Mortality of persons with epilepsy accounted for 17·1% (95%CI:14·0-20·7%) of the overall number of deaths in the population.

Interpretation In onchocerciasis-endemic areas with high prevalence of epilepsy, strengthening onchocerciasis elimination interventions can decrease the incidence of epilepsy, including NS. Additional efforts are needed in Maridi, where epilepsy is a major cause of mortality, to increase CDTi coverage and sustain blackfly control.

ELIGIBILITY:
Inclusion Criteria:

* entire population of selected villages in Maridi County

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study was conducted in 44 villages from eight study areas in the central area of Maridi County: Hai-Gabat, Hai-Matara, Hai-Tarawa, Kazana-1, Kazana-2, Kwanga, Mudubai and Nagbaka.
Sampling Method: Probability Sample
Enrollment: 17000 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-02-19 (Actual)

PRIMARY OUTCOMES:
epilepsy incidence | 4 years
  Incidence of epilepsy including nodding syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Jane Carter, MD, Principal Investigator — Amref Health Africa
Locations (1):
- Amref Health Africa, Juba, Central, South Sudan

IPD SHARING:
Plan to Share IPD: No
After de-identification (text, tables, figures, and appendices), all individual participant data that underlie the results reported in this article will be made available immediately and indefinitely via the Zenodo repository following publication for anyone who wishes to access the data for any purpose.